CLINICAL TRIAL: NCT04727866
Title: Motor Cortex Plus Spinal Cord Stimulation for Chronic Cervical Spinal Cord Injury
Brief Title: Brain Plus Spinal Stimulation for Cervical SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Collaborators: New York State Department of Health (Other Government)
Responsible Party: Principal Investigator, Noam Y. Harel, Staff Physician, Bronx VA Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HAR-19-57; C31291 (Other Grant/Funding Number: New York State Department of Health)
Record Dates: First submitted 2020-11-13; First posted 2021-01-27 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Spinal Cord Injuries; Spinal Cord Injury at C5-C7 Level; Tetraplegia/Tetraparesis
Keywords: transcranial magnetic stimulation; spinal direct current stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Rostral tsDCS (Experimental): DCS cathode over ~C3-C5 posteriorly, anode over ~C5-T1 anteriorly
  Interventions: Device: transcutaneous spinal direct current stimulation (tsDCS) - rostral; Device: intermittent theta burst stimulation (iTBS)
- Caudal tsDCS (Experimental): DCS cathode over ~T1-T4 posteriorly, anode over ~C5-T1 anteriorly
  Interventions: Device: transcutaneous spinal direct current stimulation (tsDCS) - caudal; Device: intermittent theta burst stimulation (iTBS)
- Coronal tsDCS (Experimental): DCS cathode over C5-C7 transverse process on target side, anode over C5-C7 transverse process on non-target side.
  Interventions: Device: transcutaneous spinal direct current stimulation (tsDCS) - coronal

INTERVENTIONS:
Device: transcutaneous spinal direct current stimulation (tsDCS) - coronal — 20 minutes of tsDCS will be delivered at 66% of maximum tolerated intensity with cathode over C5-C7 transverse process on target side, anode over C5-C7 transverse process on non-target side.
  Arms: Coronal tsDCS
Device: transcutaneous spinal direct current stimulation (tsDCS) - caudal — 20 minutes of tsDCS will be delivered at 66% of maximum tolerated intensity with DCS cathode over ~T1-T4 posteriorly, anode over ~C5-T1 anteriorly
  Arms: Caudal tsDCS
Device: transcutaneous spinal direct current stimulation (tsDCS) - rostral — 20 minutes of tsDCS will be delivered at 66% of maximum tolerated intensity with DCS cathode over ~C3-C5 posteriorly, anode over ~C5-T1 anteriorly
  Arms: Rostral tsDCS
Device: intermittent theta burst stimulation (iTBS) — 3 minutes of iTBS (a form of repetitive TMS) will be delivered during a 5-minute interval of DCS
  Arms: Caudal tsDCS; Rostral tsDCS

SUMMARY:
The goal of this project is to strengthen residual corticospinal tract (CST) connections after partial injury using combined motor cortex and spinal cord stimulation to improve arm and hand function after spinal cord injury (SCI).

To do this, the investigators will test the combination of transcranial magnetic stimulation (TMS) with transcutaneous spinal direct current stimulation (tsDCS) in individuals with chronic cervical SCI.

DETAILED DESCRIPTION:
For people with cervical SCI, regaining hand function is their highest priority. Most SCIs are motor incomplete, and even when complete, there is often significant amounts of spared spinal cord white matter. The goal of this project is to strengthen residual corticospinal tract (CST) connections after partial injury using combined motor cortex and spinal cord stimulation to improve arm and hand function.

The team's research in rats, which has been refined in over a decade of study, demonstrates that brain and spinal cord stimulation fully restores motor skills in rats after CST injury. Most significant for the population of people living with SCI, this approach is effective in the chronic phase of injury.

Recently, the investigators translated this electrical stimulation protocol into one that can be rapidly translated into people using non-invasive techniques. In rats, combined electrical intermittent theta burst stimulation (iTBS) of motor cortex with transcutaneous spinal direct current stimulation (tsDCS) activates the cervical spinal cord. This protocol, which is administered only 30 minutes a day for 10 days, causes large-scale sprouting of CST connections and full recovery of forelimb function. Thus, by combining brain and spinal cord electrical stimulation in rodents with corticospinal system injury durable CST axonal sprouting, strengthening of CST connections, and recovery is achieved.

In this proposal, the investigators intend to bring this promising therapeutic approach to humans with cervical SCI. The team will study people with chronic, motor incomplete, SCI to test the safety and feasibility of this approach. The investigators' approach is non-invasive and, if shown to be effective, can be rapidly integrated into current clinical practice to help restore hand function in people with chronic SCI.

Each subject will undergo four stimulation sessions of 4 hours or less. Outcomes focus on safety and neurophysiological transmission. The first session is used to determine the target muscle, optimal scalp site for TMS stimulation, assess cervical tsDCS tolerability, and measure maximal contraction force of the fingers, wrist, and elbow. The second through fourth sessions will assess the acute tolerability and effects of tsDCS with different intensities and electrode configurations in a randomized order. Each session will test a different electrode configuration and will be divided into two stages. The first stage will randomly deliver three 5-minute blocks of tsDCS at different randomized intensities (100%, 66% and 0% (sham) of tolerated intensity, as determined in Session 1) and assess changes in corticospinal and spinal excitability in response to TMS and peripheral nerve stimulation (PNS) of the target muscle. The second stage will assess the acute effects of 20-minutes of tsDCS delivered at two thirds the maximal tolerability on TMS- and PNS-evoked responses and performance of a motor task. Safety and tolerability will be closely monitored at all times.

ELIGIBILITY:
Inclusion Criteria:

Able-bodied participants

1. Age between 18 and 75 years;
2. No known central or peripheral neurological disease or injury.

SCI participants

1. Age between 18 and 75 years;
2. Chronic (> 12 months) SCI between neurological levels C1-C8;
3. Score of 2, 3, or 4 (out of 5) on manual muscle testing of elbow flexion, wrist extension, wrist flexion, finger extension, finger flexion, or finger abduction in left or right hand;

Exclusion Criteria:

1. Multiple spinal cord lesions;
2. History of seizures;
3. Ventilator dependence or patent tracheostomy site;
4. Use of medications that significantly lower seizure threshold, such as amphetamines, neuroleptics, dalfampridine, and bupropion;
5. History of stroke, brain tumor, or brain abscess;
6. History of moderate or severe head trauma (loss of consciousness for greater than one hour or evidence of brain contusion or hemorrhage or depressed skull fracture on prior imaging);
7. History of implanted brain/spine/nerve stimulators, aneurysm clips, ferromagnetic metallic implants, or cardiac pacemaker/defibrillator;
8. Significant coronary artery or cardiac conduction disease;
9. Recent history (within past 6 months) of recurrent autonomic dysreflexia, defined as a syndrome of sudden rise in systolic pressure greater than 20 mm Hg or diastolic pressure greater than 10 mm Hg, without rise in heart rate, accompanied by symptoms such as headache, facial flushing, sweating, nasal congestion, and blurry vision (this will be closely monitored during all screening and testing procedures);
10. History of bipolar disorder;
11. History of suicide attempt;
12. Active psychosis;
13. Heavy alcohol consumption (greater than equivalent of 5 oz of liquor) within previous 48 hours;
14. Open skin lesions over the face, neck, shoulders, or arms;
15. Pregnancy;
16. Unsuitable for study participation as determined by study physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-13 (Actual)

PRIMARY OUTCOMES:
Motor evoked potential (MEP) amplitudes | Change immediately after procedure
  Response to transcranial magnetic stimulation in hand and forearm muscles

SECONDARY OUTCOMES:
H-reflex amplitudes | Change immediately after procedure
  Response to peripheral nerve stimulation in extensor and flexor carpi radialis
Muscle dynamometry | Change immediately after procedure
  Pinch and wrist extension force will be measured using dynamometry
Intracortical inhibition and facilitation | Change immediately after procedure
  Change in MEP amplitude when subthreshold conditioning pulses delivered at varying interstimulus intervals

CONTACTS AND LOCATIONS:
Overall Officials: Noam Y Harel, MD, PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters Veterans Affairs Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified, individual-level data will be deposited to appropriate public repositories, such as Open Data Commons for Spinal Cord Injury (https://scicrunch.org/odc-sci), Figshare, or others.
  This will allow more powerful meta-analysis of disparate smaller studies, a need which is even more urgent in neurorehabilitation than in other fields that are more amenable to large drug studies.
Supporting Information: Study Protocol, SAP
Time Frame: Within 6 months of manuscript preparation.
Access Criteria: Individually identifiable data will be shared pursuant to valid HIPAA Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions described in the authorization and consent.
  A Data Use Agreement (DUA) will indicate adherence to any applicable Informed Consent provisions, and prohibits the recipient from identifying or re-identifying any individual whose data are included in the dataset.